CLINICAL TRIAL: NCT03421431
Title: A Phase 2 Dose Ranging, Randomized, Double Blind, and Placebo-Controlled Study Evaluating the Safety, Tolerability, Pharmacokinetics and Efficacy of EDP-305 in Subjects With Non-Alcoholic Steatohepatitis (NASH)
Brief Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics and Efficacy of EDP-305 in Subjects With Non-Alcoholic Steatohepatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Enanta Pharmaceuticals, Inc (Industry)
Collaborators: ICON Clinical Research (Industry); Triangle Biostatistics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EDP 305-101
Record Dates: First submitted 2018-01-29; First posted 2018-02-05 (Actual); Results first posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-08

CONDITIONS: Non-Alcoholic Steatohepatitis
Keywords: NASH; Non-Alcoholic Steatohepatitis (NASH)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- EDP-305 Dose 1 (Experimental): Subjects will take 2 tablets once a day orally for 12 weeks
  Interventions: Drug: EDP-305 Dose 1
- EDP-305 Dose 2 (Experimental): Subjects will take 2 tablets once a day orally for 12 weeks
  Interventions: Drug: EDP-305 Dose 2
- Placebo (Placebo Comparator): Subjects will take 2 tablets once a day orally for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EDP-305 Dose 1 — Two tablets daily for 12 weeks
  Arms: EDP-305 Dose 1
Drug: EDP-305 Dose 2 — Two tablets daily for 12 weeks
  Arms: EDP-305 Dose 2
Drug: Placebo — Two tablets daily for 12 weeks
  Arms: Placebo

SUMMARY:
A randomized, double-blind study to assess the safety, tolerability, PK and efficacy of EDP-305 in subjects with Non-Alcoholic Steatohepatitis

ELIGIBILITY:
Inclusion Criteria:

* An informed consent document must be signed and dated by the subject
* Male and female subjects of any ethnic origin between the ages of 18 and 75 years, inclusive
* Male or female with presence of NASH by:

  * Histologic evidence on a historical liver biopsy within 24 months of Screening consistent with NASH with fibrosis (no cirrhosis), and elevated ALT at Screening AND Screening MRI PDFF with >8 % steatosis OR
  * Phenotypic diagnosis of NASH based on elevated ALT and diagnosis of T2DM or pre-diabetes AND Screening MRI PDFF with >8 % steatosis
* Body mass index (BMI) >25 kg/m2; for Asian-Americans, BMI >23 kg/m2
* Female subjects of childbearing potential must agree to use two effective methods of contraception from the date of Screening until 90 days after the last dose of EDP-305.
* Subject must be willing and able to adhere to the assessments, visit schedules, prohibitions and restrictions, as described in this protocol

Exclusion Criteria:

* Laboratory Screening Results:

  * Total bilirubin > ULN (normal range 0.2-1.2 mg/dL)
  * Total white blood cells (WBC) <3,000 cells/mm3
  * Absolute neutrophil count (ANC) <1,500 cells/mm3
  * Platelet count <140,000/mm3
  * Prothrombin time (international normalized ratio, INR) > 1.2
  * Creatine kinase above the upper limit of normal (ULN) except when in relation with intense exercise
  * Serum creatinine >2 mg/dL or creatinine clearance <60 ml/min (based on Cockroft Gault method)
* Known history of alpha-1-antitrypsin deficiency
* Use of an experimental treatment for NASH within the past 6 months
* Use of immunosuppressant (eg, corticosteroids) for more than 2 weeks in duration within 1 year prior to Screening and during the course of the study
* Use of experimental or unapproved drugs within a year of Screening
* Any other condition(s) (including cardiovascular diseases) that would compromise the safety of the subject or compromise the quality of the clinical study, as judged by the Principal Investigator (PI)
* Pregnant or nursing females
* Recipients of liver or other organ transplantation or anticipated need for orthotropic organ transplantation in one year as determined by a Model for End-Stage Liver Disease (MELD) Score ≥ 15
* Clinical suspicion of advanced liver disease or cirrhosis
* Coexisting liver or biliary diseases, such as primary sclerosing cholangitis (PSC), choledocholithiasis, acute or chronic hepatitis, autoimmune hepatitis, alcoholic liver disease, acute infection of bile duct system or gall bladder, history of gastrointestinal bleeding (secondary to portal hypertension), cirrhosis
* Suspicion of cancer (eg, liver cancer) with the exception of basal cell carcinoma that has been resected
* Cirrhosis with or without complications, including history or presence of: spontaneous bacterial peritonitis, hepatocellular carcinoma, bilirubin > 2xULN
* Hepatorenal syndrome (type I or II) or Screening serum creatinine > 2 mg/dL (178 μmol/L)
* Prior variceal hemorrhage, uncontrolled encephalopathy, Child-Pugh Class A, B, and C, esophageal varices, or refractory ascites within the previous 6 months of Screening (defined as date informed consent signed)
* Any condition possibly affecting drug absorption (eg, gastrectomy <3 years prior to Screening)
* Subject has received an investigational agent or vaccine within 30 days, or a biological product within 3 months or 5 elimination half-lives (whichever is longer) prior to the planned intake of study drug. NOTE: Flu vaccine will be allowed upon Medical Monitor's approval
* Use of a new statin regimen from Screening and throughout study duration. NOTE: Subjects on a stable dose of statins for at least three months prior to Screening are allowed. No dose modification during the study will be allowed.
* Current use of fibrates. Note: Subjects who discontinued fibrates for at least 3 months before Screening can participate
* Clinically significant history of drug sensitivity or allergy, as determined by the PI
* Uncontrolled diabetes mellitus (ie, HbA1c ≥9% or higher) 60 days prior to Day 1
* Subjects with contraindications to MRI imaging, or not being able to have the MRI performed

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2019-06-14 (Actual); Study Completion 2019-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Adda, MD, Study Director — Enanta Pharmaceuticals, Inc
Locations (82):
- United States (70):
  - Radiant Research Incorporated, Chandler, Arizona
  - Central Arizona Medical Associates, Mesa, Arizona
  - Mayo Clinic Specialty Building, Phoenix, Arizona
  - Anaheim Clinical Trials, Anaheim, California
  - estudy site - Chula Vista, Chula Vista, California
  - Southern California Research Center, Coronado, California
  - Fresno Clinical Research Center (FCRC), Fresno, California
  - UCSD Altman Clinical and Translational Research Institute, La Jolla, California
  - Clinical Trials Research, Lincoln, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - National Research Institute, Los Angeles, California
  - Catalina Research Institute, LLC, Montclair, California
  - Inland Empire Liver Foundation, Rialto, California
  - Southern California Transplantation Institute Research Foundation, San Clemente, California
  - Precision Research Institute, San Diego, California
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Clinical Research Advantage, Inc. / Colorado Springs Family Practice, Colorado Springs, Colorado
  - South Denver Gastroenterology,P.C., Englewood, Colorado
  - Avail Clinical Research, LLC, DeLand, Florida
  - Fleming Island Center for Clinical Research, Fleming Island, Florida
  - Westside Center for Clinical Research, Jacksonville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Jacksonville Center for Endoscopy - Southside ; Borland Groover Clinic, Jacksonville, Florida
  - Precision Clinical Research, LLC., Lauderdale Lakes, Florida
  - Homestead Medical Research, Miami, Florida
  - Research Associates of South Florida, LLC, Miami, Florida
  - Florida Advanced Medical Research, Inc., Miami, Florida
  - Ocean Blue Medical Research Center, Inc, Miami Springs, Florida
  - Clinical Neuroscience Solutions Inc., Orlando, Florida
  - Advanced Gastroenterology Associates, LLC, Palm Harbor, Florida
  - Piedmont Atlanta Hospital, Atlanta, Georgia
  - Gastrointestinal Specialists Of Georgia, Marietta, Georgia
  - Feinberg School of Medicine Northwestern University, Chicago, Illinois
  - Midwest Institute For Clinical Research, Indianapolis, Indiana
  - WestGlen Gastrointestinal Consultants, PA, Shawnee Mission, Kansas
  - Oshsner Clinic Foundation, New Orleans, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Digestive Disease Associates, PA, Catonsville, Maryland
  - University of Michigan Health System, Ann Arbor, Michigan
  - Kansas City Research Institute, Kansas City, Missouri
  - Saint Louis University, St Louis, Missouri
  - AGA Clinical Research Associates, LLC, Egg Harbor, New Jersey
  - Northwell Health Inc., Manhasset, New York
  - NYU Langone Medical Center - The Center for Musculoskeletal Care (CMC), New York, New York
  - Weill Cornell Medical College, New York, New York
  - Carolinas Medical Center Transplant Center/Center for Liver Disease, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Carolinas Center for Liver Disease / Carolinas Health Care System, Huntersville, North Carolina
  - Sterling Research Group, Ltd., Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pittsburgh Medical Center - Center for Liver Diseases, Pittsburgh, Pennsylvania
  - University Of Tennessee Health Science Center, Memphis, Tennessee
  - Quality Medical Research, PLLC, Nashville, Tennessee
  - Texas Clinical Research Institute, Arlington, Texas
  - Texas Diabetes & Endocrinology, Austin, Texas
  - Dallas Diabetes Research Center, Dallas, Texas
  - DHAT Research Institute, Garland, Texas
  - Baylor College of Medicine - Advanced Liver Therapies, Houston, Texas
  - Texas Liver Institute, San Antonio, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Radiant Research, Inc., San Antonio, Texas
  - Wasatch Peak Family Practice/Radiant Research, Inc, Layton, Utah
  - Radiant Research, Inc., Murray, Utah
  - Gastroenterology Associates, PC, Gainesville, Virginia
  - Bon Secours St. Mary's Hospital of Richmond, Inc, Newport News, Virginia
  - The Gastroenterology Group, PC, Reston, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Swedish Medical Center-Swedish Organ Transplant and Liver Center, Seattle, Washington
  - University of Washington / Harborview Medical Center, Seattle, Washington
  - Mayo Clinic Health System - Franciscan Healthcare, La Crosse, Wisconsin
- Canada (4):
  - Aggarwal and Associates Limited, Brampton, Ontario
  - Toronto Liver Centre, Toronto, Ontario
  - Clinique de recherche Medpharmgene, Montreal, Quebec
  - Chronic Viral Illness Service McGill University Health Center/Royal Victoria, Montreal, Quebec
- France (3):
  - Hopital Pitie Salpetriere, Paris
  - CHU de Bordeaux - GH Sud - Hoital Haut Leveque, Pessac
  - CHU de Strasbourg - Nouvel Hôspital Civil, Strasbourg
- Auckland Clinical Studies Limited, Auckland, New Zealand
- Latin Clinical Trial Center, San Juan, Puerto Rico
- United Kingdom (3):
  - Addenbrookes Hospital (AH)-Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambridgeshire
  - King's College Hospital NHS Foundation, London, Greater London
  - Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ratziu V, Rinella ME, Neuschwander-Tetri BA, Lawitz E, Denham D, Kayali Z, Sheikh A, Kowdley KV, Desta T, Elkhashab M, DeGrauw J, Goodwin B, Ahmad A, Adda N. EDP-305 in patients with NASH: A phase II double-blind placebo-controlled dose-ranging study. J Hepatol. 2022 Mar;76(3):506-517. doi: 10.1016/j.jhep.2021.10.018. Epub 2021 Nov 3. PMID 34740705

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Safety or Efficacy Population consisted of all participants who received at least one dose of the study treatment. Out of 134 randomized participants, 2 participants (1 participant each in the EDP-305 2.5 mg and placebo groups) were randomized but not dosed because the participants withdrew and were not included in the Safety and Efficacy Populations.
Groups:
- Placebo: A matching placebo tablet (EDP-305 1 mg or 2.5 mg) was administered orally once daily in the morning after fasting overnight for a minimum of 8 hours for 12 weeks. The matching placebo contained all the excipients present in the EDP-305 drug product tablets with the exception of the active drug.
- EDP-305 1 mg: EDP-305 1 mg tablet was administered orally once daily in the morning after fasting overnight for a minimum of 8 hours for 12 weeks.
- EDP-305 2.5 mg: EDP-305 2.5 mg tablet was administered orally once daily in the morning after fasting overnight for a minimum of 8 hours for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | EDP-305 1 mg | EDP-305 2.5 mg
Started | 24 | 55 | 53
Completed | 18 | 49 | 39
Not Completed | 6 | 6 | 14
Not completed — Adverse Event | 2 | 1 | 12
Not completed — Lost to Follow-up | 1 | 1 | 1
Not completed — Withdrawal by Subject | 3 | 2 | 1
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Participant met Stopping Rules | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Demographics were summarized for the Safety Population, which included all the randomized participants who received at least one dose of the study treatment.
  The numbers of participants included in the Efficacy Population were same as the Safety Population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | EDP-305 1 mg | EDP-305 2.5 mg | Total
Number analyzed (Participants) | 24 | 55 | 53 | 132
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 22 | 52 | 46 | 120
  ≥65 years | 2 | 3 | 7 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 29 | 29 | 69
  Male | 13 | 26 | 24 | 63
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 1 | 7 | 3 | 11
  Black or African American | 2 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  White | 17 | 42 | 47 | 106
  Not reported | 2 | 2 | 1 | 5
  Other | 0 | 0 | 1 | 1
  Mexican | 1 | 1 | 1 | 3
  Not specified | 0 | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline (Average) in Alanine Aminotransferase (ALT) at Week 12
Description: Blood samples were collected at specific timepoints for the laboratory evaluation to assess the ALT level. Baseline refers to the average of the screening and the Day 1 values; if either the screening or Day 1 values were missing, the non-missing value was used. Mean change was defined as the mean value at Week 12 minus the mean value at baseline.
Time Frame: Baseline and Week 12
Population: Efficacy Population: included all participants who received at least one dose of the study treatment. Here "Overall Number of Participants Analyzed" = participants evaluable for this outcome measure. Only those participants with valid measurements for the outcome measure at the specified time point were reported.
Measure: Mean (Standard Deviation); unit: units per liter (U/L)
Arm/Group | Placebo | EDP-305 1 mg | EDP-305 2.5 mg
Number analyzed (Participants) | 20 | 48 | 38
units per liter (U/L) | -13.85 (18.151) | -23.76 (28.135) | -26.14 (33.328)
Statistical Analysis 1: Comparison: Placebo vs EDP-305 2.5 mg; Test type: Superiority; p = 0.0495, ANCOVA; Least Squares (LS) mean difference = 12.460, 95% CI 2-sided [0.029 to 24.891]
Statistical Analysis 2: Comparison: Placebo vs EDP-305 1 mg; Test type: Superiority; p = 0.3039, ANCOVA; LS mean difference = 6.257, 95% CI 2-sided [-5.754 to 18.268]
Statistical Analysis 3: Comparison: EDP-305 1 mg vs EDP-305 2.5 mg; Test type: Superiority; p = 0.2130, ANCOVA; LS mean difference = 6.203, 95% CI 2-sided [-3.615 to 16.021]

2. Secondary Outcome: Mean Change From Baseline in Percentage of Fat in the Liver as Assessed by Magnetic Resonance Imaging - Proton Density Fat Fraction (MRI-PDFF) at Week 12
Description: The liver fat percentage was assessed by MRI-PDFF, which is an established method that enables the quantification of fat content in the liver; the value of liver fat is expressed in percentage and ranges from 0 to 100% with higher values representing higher liver fat level. Baseline refers to the last non-missing value collected prior to the first dose of study treatment. Mean change was defined as the mean value at Week 12 minus the mean value at baseline.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of fat
Arm/Group | Placebo | EDP-305 1 mg | EDP-305 2.5 mg
Number analyzed (Participants) | 20 | 51 | 49
percentage of fat | -2.842 (4.4687) | -3.759 (5.1600) | -6.428 (7.2586)
Statistical Analysis 1: Comparison: Placebo vs EDP-305 2.5 mg; Test type: Superiority; p = 0.0009, ANCOVA; LS mean difference = 4.717, 95% CI 2-sided [1.980 to 7.455]
Statistical Analysis 2: Comparison: Placebo vs EDP-305 1 mg; Test type: Superiority; p = 0.4946, ANCOVA; LS mean difference = 0.934, 95% CI 2-sided [-1.766 to 3.635]
Statistical Analysis 3: Comparison: EDP-305 1 mg vs EDP-305 2.5 mg; Test type: Superiority; p = 0.0005, ANCOVA; LS mean difference = 3.783, 95% CI 2-sided [1.708 to 5.858]

3. Secondary Outcome: Mean Change From Baseline in Aspartate Aminotransferase to Platelet Ratio Index (APRI) at Week 12
Description: Blood samples were collected at specific timepoints for the laboratory evaluation to assess the aspartate aminotransferase (AST) level and platelet count. Baseline refers to the last non-missing value collected prior to the first dose of study treatment. The APRI score (AST to platelet ratio index) is an index comprised of biochemical values and is used to determine the degree of hepatic fibrosis. APRI is calculated from the level of AST measured in a blood test (international units per liter [IU/L]) and platelet count (10^9/L) according to the following formula:
  APRI = ([AST value in IU/L / upper limit of the normal range of AST] / [platelet count in 10^9/L]) × 100.
  In general, APRI scores range from 0 to >2.0, where scores <0.5 indicate no significant fibrosis, scores >1.5 indicate significant fibrosis, and scores >2.0 have been shown to be best correlated with the presence of cirrhosis. Mean change was defined as the mean value at Week 12 minus the mean value at baseline.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Placebo | EDP-305 1 mg | EDP-305 2.5 mg
Number analyzed (Participants) | 17 | 44 | 35
ratio | -0.180 (0.3462) | -0.107 (0.3396) | -0.194 (0.3533)
Statistical Analysis 1: Comparison: Placebo vs EDP-305 2.5 mg; Test type: Superiority; p = 0.2756, ANCOVA; LS mean difference = 0.076, 95% CI 2-sided [-0.062 to 0.214]
Statistical Analysis 2: Comparison: Placebo vs EDP-305 1 mg; Test type: Superiority; p = 0.9686, ANCOVA; LS mean difference = -0.003, 95% CI 2-sided [-0.136 to 0.131]
Statistical Analysis 3: Comparison: EDP-305 1 mg vs EDP-305 2.5 mg; Test type: Superiority; p = 0.1406, ANCOVA; LS mean difference = 0.079, 95% CI 2-sided [-0.026 to 0.184]

4. Secondary Outcome: Mean Change From Baseline in Triglycerides (TG) at Week 12
Description: Blood samples were collected at specific timepoints for the laboratory evaluation to assess the TG level. Baseline refers to the last non-missing value collected prior to the first dose of study treatment. Mean change was defined as the mean value at Week 12 minus the mean value at baseline.
Time Frame: Baseline and Week 12
Population: Efficacy Population: included all participants who received at least one dose of the study treatment. Here "Overall Number of Participants Analyzed"= participants evaluable for this outcome measure. Only those participants with valid measurements for the outcome measure at the specified time point were reported.
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Placebo | EDP-305 1 mg | EDP-305 2.5 mg
Number analyzed (Participants) | 20 | 48 | 38
millimoles per liter (mmol/L) | -0.151 (0.8529) | -0.366 (1.5858) | 0.129 (1.1088)
Statistical Analysis 1: Comparison: Placebo vs EDP-305 2.5 mg; Test type: Superiority; p = 0.6130, ANCOVA; LS mean difference = -0.125, 95% CI 2-sided [-0.613 to 0.363]
Statistical Analysis 2: Comparison: Placebo vs EDP-305 1 mg; Test type: Superiority; p = 0.8366, ANCOVA; LS mean difference = -0.049, 95% CI 2-sided [-0.521 to 0.423]
Statistical Analysis 3: Comparison: EDP-305 1 mg vs EDP-305 2.5 mg; Test type: Superiority; p = 0.7015, ANCOVA; LS mean difference = -0.076, 95% CI 2-sided [-0.466 to 0.315]

5. Secondary Outcome: Mean Change From Baseline in Total Cholesterol at Week 12
Description: Blood samples were collected at specific timepoints for the laboratory evaluation to assess the total cholesterol level. Baseline refers to the last non-missing value collected prior to the first dose of study treatment. Mean change was defined as the mean value at Week 12 minus the mean value at baseline.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | EDP-305 1 mg | EDP-305 2.5 mg
Number analyzed (Participants) | 20 | 49 | 38
mmol/L | -0.175 (0.6879) | 0.046 (0.6697) | -0.003 (1.0046)
Statistical Analysis 1: Comparison: Placebo vs EDP-305 2.5 mg; Test type: Superiority; p = 0.3875, ANCOVA; LS mean difference = -0.186, 95% CI 2-sided [-0.613 to 0.240]
Statistical Analysis 2: Comparison: Placebo vs EDP-305 1 mg; Test type: Superiority; p = 0.2331, ANCOVA; LS mean difference = -0.248, 95% CI 2-sided [-0.657 to 0.162]
Statistical Analysis 3: Comparison: EDP-305 1 mg vs EDP-305 2.5 mg; Test type: Superiority; p = 0.7164, ANCOVA; LS mean difference = 0.061, 95% CI 2-sided [-0.272 to 0.395]

6. Secondary Outcome: Mean Change From Baseline in High-Density Lipoprotein Cholesterol (HDL-C) at Week 12
Description: Blood samples were collected at specific timepoints for the laboratory evaluation to assess the HDL-C level. Baseline refers to the last non-missing value collected prior to the first dose of study treatment. Mean change was defined as the mean value at Week 12 minus the mean value at baseline.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | EDP-305 1 mg | EDP-305 2.5 mg
Number analyzed (Participants) | 20 | 49 | 38
mmol/L | 0.008 (0.1279) | -0.058 (0.1670) | -0.210 (0.2708)
Statistical Analysis 1: Comparison: Placebo vs EDP-305 2.5 mg; Test type: Superiority; p < 0.0001, ANCOVA; LS mean difference = 0.210, 95% CI 2-sided [0.110 to 0.311]
Statistical Analysis 2: Comparison: Placebo vs EDP-305 1 mg; Test type: Superiority; p = 0.3480, ANCOVA; LS mean difference = 0.046, 95% CI 2-sided [-0.051 to 0.143]
Statistical Analysis 3: Comparison: EDP-305 1 mg vs EDP-305 2.5 mg; Test type: Superiority; p < 0.0001, ANCOVA; LS mean difference = 0.164, 95% CI 2-sided [0.085 to 0.243]

7. Secondary Outcome: Mean Change From Baseline in Low-Density Lipoprotein Cholesterol (LDL-C) at Week 12
Description: Blood samples were collected at specific timepoints for the laboratory evaluation to assess the LDL-C level. Baseline refers to the last non-missing value collected prior to the first dose of study treatment. Mean change was defined as the mean value at Week 12 minus the mean value at baseline.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | EDP-305 1 mg | EDP-305 2.5 mg
Number analyzed (Participants) | 20 | 44 | 37
mmol/L | -0.112 (0.6431) | 0.129 (0.5099) | 0.151 (0.8157)
Statistical Analysis 1: Comparison: Placebo vs EDP-305 2.5 mg; Test type: Superiority; p = 0.0897, ANCOVA; LS mean difference = -0.299, 95% CI 2-sided [-0.645 to 0.047]
Statistical Analysis 2: Comparison: Placebo vs EDP-305 1 mg; Test type: Superiority; p = 0.1411, ANCOVA; LS mean difference = -0.251, 95% CI 2-sided [-0.586 to 0.085]
Statistical Analysis 3: Comparison: EDP-305 1 mg vs EDP-305 2.5 mg; Test type: Superiority; p = 0.7330, ANCOVA; LS mean difference = -0.048, 95% CI 2-sided [-0.326 to 0.230]

8. Secondary Outcome: Mean Change From Baseline in Adiponectin at Week 12
Description: Blood samples were collected at specific timepoints for the laboratory evaluation to assess the adiponectin level. Baseline refers to the last non-missing value collected prior to the first dose of study treatment. Mean change was defined as the mean value at Week 12 minus the mean value at baseline.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Placebo | EDP-305 1 mg | EDP-305 2.5 mg
Number analyzed (Participants) | 20 | 48 | 38
nanogram per milliliter (ng/mL) | 319.16 (689.387) | 17.94 (828.494) | 522.00 (2649.701)
Statistical Analysis 1: Comparison: Placebo vs EDP-305 2.5 mg; Test type: Superiority; p = 0.9143, ANCOVA; LS mean difference = 51.873, 95% CI 2-sided [-901.574 to 1005.320]
Statistical Analysis 2: Comparison: Placebo vs EDP-305 1 mg; Test type: Superiority; p = 0.3718, ANCOVA; LS mean difference = 404.168, 95% CI 2-sided [-489.519 to 1297.854]
Statistical Analysis 3: Comparison: EDP-305 1 mg vs EDP-305 2.5 mg; Test type: Superiority; p = 0.3466, ANCOVA; LS mean difference = -352.295, 95% CI 2-sided [-1091.308 to 386.719]

9. Secondary Outcome: Mean Change From Baseline in Apolipoproteins A1 (ApoA-1) at Week 12
Description: Blood samples were collected at specific timepoints for the laboratory evaluation to assess the ApoA-1 level. Baseline refers to the last non-missing value collected prior to the first dose of study treatment. Mean change was defined as the mean value at Week 12 minus the mean value at baseline.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: proteins*10^9/L
Arm/Group | Placebo | EDP-305 1 mg | EDP-305 2.5 mg
Number analyzed (Participants) | 20 | 49 | 38
proteins*10^9/L | -0.074 (0.1514) | -0.107 (0.1671) | -0.226 (0.2197)
Statistical Analysis 1: Comparison: Placebo vs EDP-305 2.5 mg; Test type: Superiority; p = 0.0003, ANCOVA; LS mean difference = 0.173, 95% CI 2-sided [0.081 to 0.264]
Statistical Analysis 2: Comparison: Placebo vs EDP-305 1 mg; Test type: Superiority; p = 0.5685, ANCOVA; LS mean difference = 0.025, 95% CI 2-sided [-0.062 to 0.113]
Statistical Analysis 3: Comparison: EDP-305 1 mg vs EDP-305 2.5 mg; Test type: Superiority; p < 0.0001, ANCOVA; LS mean difference = 0.147, 95% CI 2-sided [0.075 to 0.219]

10. Secondary Outcome: Mean Change From Baseline in Apolipoproteins B (ApoB) at Week 12
Description: Blood samples were collected at specific timepoints for the laboratory evaluation to assess the ApoB level. Baseline refers to the last non-missing value collected prior to the first dose of study treatment. Mean change was defined as the mean value at Week 12 minus the mean value at baseline.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: proteins*10^9/L
Arm/Group | Placebo | EDP-305 1 mg | EDP-305 2.5 mg
Number analyzed (Participants) | 20 | 49 | 38
proteins*10^9/L | -0.028 (0.1687) | 0.040 (0.1781) | 0.099 (0.2898)
Statistical Analysis 1: Comparison: Placebo vs EDP-305 2.5 mg; Test type: Superiority; p = 0.0282, ANCOVA; LS mean difference = -0.133, 95% CI 2-sided [-0.252 to -0.015]
Statistical Analysis 2: Comparison: Placebo vs EDP-305 1 mg; Test type: Superiority; p = 0.2412, ANCOVA; LS mean difference = -0.068, 95% CI 2-sided [-0.182 to 0.046]
Statistical Analysis 3: Comparison: EDP-305 1 mg vs EDP-305 2.5 mg; Test type: Superiority; p = 0.1649, ANCOVA; LS mean difference = -0.066, 95% CI 2-sided [-0.158 to 0.027]

11. Secondary Outcome: Mean Change From Baseline in Apolipoproteins C3 (ApoC3) at Week 12
Description: Blood samples were collected at specific timepoints for the laboratory evaluation to assess the ApoC3 level. Baseline refers to the last non-missing value collected prior to the first dose of study treatment. Mean change was defined as the mean value at Week 12 minus the mean value at baseline.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: proteins*10^9/L
Arm/Group | Placebo | EDP-305 1 mg | EDP-305 2.5 mg
Number analyzed (Participants) | 20 | 49 | 38
proteins*10^9/L | -0.0094 (0.04388) | -0.0167 (0.03918) | -0.0122 (0.05721)
Statistical Analysis 1: Comparison: Placebo vs EDP-305 2.5 mg; Test type: Superiority; p = 0.4357, ANCOVA; LS mean difference = 0.009, 95% CI 2-sided [-0.014 to 0.032]
Statistical Analysis 2: Comparison: Placebo vs EDP-305 1 mg; Test type: Superiority; p = 0.8989, ANCOVA; LS mean difference = 0.001, 95% CI 2-sided [-0.021 to 0.023]
Statistical Analysis 3: Comparison: EDP-305 1 mg vs EDP-305 2.5 mg; Test type: Superiority; p = 0.4120, ANCOVA; LS mean difference = 0.008, 95% CI 2-sided [-0.011 to 0.026]

12. Secondary Outcome: Mean Change From Baseline in Fasting Blood Glucose at Week 12
Description: Blood samples were collected at specific timepoints for the laboratory evaluation to assess the fasting glucose level. Baseline refers to the last non-missing value collected prior to the first dose of study treatment. Mean change was defined as the mean value at Week 12 minus the mean value at baseline.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | EDP-305 1 mg | EDP-305 2.5 mg
Number analyzed (Participants) | 20 | 48 | 38
mmol/L | -0.11 (2.130) | 0.48 (1.847) | 1.68 (3.396)
Statistical Analysis 1: Comparison: Placebo vs EDP-305 2.5 mg; Test type: Superiority; p = 0.0134, ANCOVA; LS mean difference = -1.731, 95% CI 2-sided [-3.095 to -0.368]
Statistical Analysis 2: Comparison: Placebo vs EDP-305 1 mg; Test type: Superiority; p = 0.6263, ANCOVA; LS mean difference = -0.327, 95% CI 2-sided [-1.656 to 1.001]
Statistical Analysis 3: Comparison: EDP-305 1 mg vs EDP-305 2.5 mg; Test type: Superiority; p = 0.0115, ANCOVA; LS mean difference = -1.404, 95% CI 2-sided [-2.487 to -0.322]

13. Secondary Outcome: Mean Change From Baseline in Fasting Insulin at Week 12
Description: Blood samples were collected at specific timepoints for the laboratory evaluation to assess the fasting insulin (in micro International units per milliliter [μIU/mL]). Baseline refers to the last non-missing value collected prior to the first dose of study treatment. Mean change was defined as the mean value at Week 12 minus the mean value at baseline.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μIU/mL
Arm/Group | Placebo | EDP-305 1 mg | EDP-305 2.5 mg
Number analyzed (Participants) | 20 | 47 | 38
μIU/mL | -0.688 (9.2808) | 2.528 (14.6947) | -5.635 (52.7637)
Statistical Analysis 1: Comparison: Placebo vs EDP-305 2.5 mg; Test type: Superiority; p = 0.4608, ANCOVA; LS mean difference = -3.723, 95% CI 2-sided [-13.700 to 6.253]
Statistical Analysis 2: Comparison: Placebo vs EDP-305 1 mg; Test type: Superiority; p = 0.6238, ANCOVA; LS mean difference = -2.377, 95% CI 2-sided [-11.962 to 7.207]
Statistical Analysis 3: Comparison: EDP-305 1 mg vs EDP-305 2.5 mg; Test type: Superiority; p = 0.7367, ANCOVA; LS mean difference = -1.346, 95% CI 2-sided [-9.268 to 6.576]

14. Secondary Outcome: Mean Change From Baseline in Homeostasis Model Assessment (HOMA) Index for Nondiabetic Participants at Week 12
Description: Blood samples were collected at specific timepoints for the laboratory evaluation; from the results of fasting glucose and insulin, an insulin resistance (IR) was estimated for the nondiabetic participants using the HOMA-IR computer algorithm. A higher HOMA-IR indicates a higher degree of insulin resistance. Participants who were not considered as having type 2 diabetes mellitus (T2DM) were identified as nondiabetic. Baseline refers to the last non-missing value collected prior to the first dose of study treatment. Mean change was defined as the mean value at Week 12 minus the mean value at baseline.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | EDP-305 1 mg | EDP-305 2.5 mg
Number analyzed (Participants) | 3 | 11 | 13
units on a scale | 0.587 (2.0088) | 0.192 (2.7180) | -6.474 (24.9369)
Statistical Analysis 1: Comparison: Placebo vs EDP-305 2.5 mg; Test type: Superiority; p = 0.8302, ANCOVA; LS mean difference = -0.407, 95% CI 2-sided [-4.287 to 3.474]
Statistical Analysis 2: Comparison: Placebo vs EDP-305 1 mg; Test type: Superiority; p = 0.5053, ANCOVA; LS mean difference = -1.280, 95% CI 2-sided [-5.192 to 2.632]
Statistical Analysis 3: Comparison: EDP-305 1 mg vs EDP-305 2.5 mg; Test type: Superiority; p = 0.4760, ANCOVA; LS mean difference = 0.873, 95% CI 2-sided [-1.620 to 3.366]

15. Secondary Outcome: Mean Change From Baseline in HOMA Index for Diabetic Participants at Week 12
Description: Blood samples were collected at specific timepoints for the laboratory evaluation; from the results of fasting glucose and insulin, an insulin resistance (IR) was estimated for the nondiabetic participants using the HOMA-IR computer algorithm. A higher HOMA-IR indicates a higher degree of insulin resistance. Participants who were considered as having T2DM were identified as diabetic. Baseline refers to the last non-missing value collected prior to the first dose of study treatment. Mean change was defined as the mean value at Week 12 minus the mean value at baseline.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | EDP-305 1 mg | EDP-305 2.5 mg
Number analyzed (Participants) | 17 | 35 | 25
units on a scale | -0.493 (6.2624) | 2.088 (6.6114) | 5.059 (15.0113)
Statistical Analysis 1: Comparison: Placebo vs EDP-305 2.5 mg; Test type: Superiority; p = 0.0639, ANCOVA; LS mean difference = -5.910, 95% CI 2-sided [-12.171 to 0.351]
Statistical Analysis 2: Comparison: Placebo vs EDP-305 1 mg; Test type: Superiority; p = 0.4884, ANCOVA; LS mean difference = -2.064, 95% CI 2-sided [-7.971 to 3.843]
Statistical Analysis 3: Comparison: EDP-305 1 mg vs EDP-305 2.5 mg; Test type: Superiority; p = 0.1532, ANCOVA; LS mean difference = -3.846, 95% CI 2-sided [-9.156 to 1.464]

16. Secondary Outcome: Mean Change From Baseline in Glycated Hemoglobin (HbA1c) in Participants With T2DM at Week 12
Description: Blood samples were collected at specific timepoints for the laboratory evaluation to assess the HbA1c. Baseline refers to the last non-missing value collected prior to the first dose of study treatment. Mean change was defined as the mean value at Week 12 minus the mean value at baseline.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin
Arm/Group | Placebo | EDP-305 1 mg | EDP-305 2.5 mg
Number analyzed (Participants) | 17 | 38 | 25
percentage of glycated hemoglobin | 0.31 (0.685) | 0.21 (0.776) | 0.76 (0.963)
Statistical Analysis 1: Comparison: Placebo vs EDP-305 2.5 mg; Test type: Superiority; p = 0.0811, ANCOVA; LS mean difference = -0.460, 95% CI 2-sided [-0.978 to 0.058]
Statistical Analysis 2: Comparison: Placebo vs EDP-305 1 mg; Test type: Superiority; p = 0.6312, ANCOVA; LS mean difference = 0.117, 95% CI 2-sided [-0.367 to 0.601]
Statistical Analysis 3: Comparison: EDP-305 1 mg vs EDP-305 2.5 mg; Test type: Superiority; p = 0.0099, ANCOVA; LS mean difference = -0.577, 95% CI 2-sided [-1.011 to -0.143]

17. Secondary Outcome: Maximum Plasma Concentration (Cmax) of EDP-305 on Day 1 and Week 12
Description: The Cmax is the maximum observed plasma concentration, which was measured for EDP-305 on Day 1 and Week 12 for the samples collected according to the intensive sampling scheme for the participants in the Pharmacokinetic (PK) Population.
Time Frame: Predose and 2, 6, and 8 hours postdose on Day 1 and on Day 84 (Week 12)
Population: PK Population: included all participants who received active study drug (EDP-305) and had any measurable plasma concentration of study drug at any timepoint. Here "Overall Number of Participants Analyzed" = participants evaluable for this outcome measure and "Number Analyzed" = participants who were evaluable for specified category.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | EDP-305 1 mg | EDP-305 2.5 mg
Number analyzed (Participants) | 54 | 52
ng/mL
  Day 1: number analyzed (Participants) | 19 | 19
  Day 1 | 11.1 (105) | 25.1 (101)
  Week 12: number analyzed (Participants) | 17 | 13
  Week 12 | 15.9 (105) | 41.1 (101)

18. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of EDP-305 on Day 1 and at Week 12
Description: The Tmax was measured for EDP-305 on Day 1 and at Week 12 for the samples collected according to the intensive sampling scheme for the participants in the PK Population.
Time Frame: Predose and 2, 6, and 8 hours postdose on Day 1 and on Day 84 (Week 12)
Population: as for outcome 17
Measure: Median (Full Range); unit: hours (h)
Arm/Group | EDP-305 1 mg | EDP-305 2.5 mg
Number analyzed (Participants) | 54 | 52
hours (h)
  Day 1: number analyzed (Participants) | 19 | 19
  Day 1 | 6.00 [2.00 to 8.07] | 6.00 [2.00 to 8.25]
  Week 12: number analyzed (Participants) | 17 | 13
  Week 12 | 6.00 [0.00 to 8.02] | 6.00 [0.00 to 8.18]

19. Secondary Outcome: Area Under the Plasma Concentration-Time Curve (AUC) From Time Zero to the Time of the Last Quantifiable Concentration (AUC[Last]) of EDP-305 on Day 1 and at Week 12
Description: AUC(last) is defined as the area under the plasma concentration-time curve from time zero to time the last quantifiable concentration, computed using the linear up/log down trapezoidal rule. AUC(last) was computed for EDP-305 on Day 1 and Week 12 for the samples collected according to the intensive sampling scheme for the participants in the PK Population.
Time Frame: Predose and 2, 6, and 8 hours postdose on Day 1 and on Day 84 (Week 12)
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | EDP-305 1 mg | EDP-305 2.5 mg
Number analyzed (Participants) | 54 | 52
hour*nanogram per milliliter (h*ng/mL)
  Day 1: number analyzed (Participants) | 19 | 19
  Day 1 | 53.6 (101) | 129 (100)
  Week 12: number analyzed (Participants) | 17 | 12
  Week 12 | 87.2 (101) | 264 (100)

20. Secondary Outcome: Cmax of EP-022571 on Day 1 and at Week 12
Description: The Cmax is the maximum observed plasma concentration, which was measured for EP-022571 (a metabolite of EDP-305) on Day 1 and Week 12 for the samples collected according to the intensive sampling scheme for the participants in the PK Population.
Time Frame: Predose and 2, 6, and 8 hours postdose on Day 1 and on Day 84 (Week 12)
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | EDP-305 1 mg | EDP-305 2.5 mg
Number analyzed (Participants) | 54 | 52
ng/mL
  Day 1: number analyzed (Participants) | 19 | 19
  Day 1 | 0.324 (983) | 0.833 (177)
  Week 12: number analyzed (Participants) | 17 | 13
  Week 12 | 0.296 (1549) | 0.787 (233)

21. Secondary Outcome: Tmax of EP-022571 on Day 1 and at Week 12
Description: The Tmax was measured for EP-022571 (a metabolite of EDP-305) on Day 1 and at Week 12 for the samples collected according to the intensive sampling scheme for the participants in the PK Population.
Time Frame: Predose and 2, 6, and 8 hours postdose on Day 1 and on Day 84 (Week 12)
Population: as for outcome 17
Measure: Median (Full Range); unit: h
Arm/Group | EDP-305 1 mg | EDP-305 2.5 mg
Number analyzed (Participants) | 54 | 52
h
  Day 1: number analyzed (Participants) | 19 | 19
  Day 1 | 6.00 [2.00 to 8.00] | 6.00 [1.93 to 8.25]
  Week 12: number analyzed (Participants) | 17 | 13
  Week 12 | 6.00 [0.00 to 8.00] | 6.00 [0.00 to 6.15]

22. Secondary Outcome: AUC(Last) of EP-022571 on Day 1 and at Week 12
Description: AUC(last) is defined as the area under the plasma concentration-time curve from time zero to time the last quantifiable concentration, computed using the linear up/log down trapezoidal rule. AUC(last) was computed for EP-022571 (a metabolite of EDP-305) on Day 1 and Week 12 for the samples collected according to the intensive sampling scheme for the participants in the PK Population.
Time Frame: Predose and 2, 6, and 8 hours postdose on Day 1 and on Day 84 (Week 12)
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | EDP-305 1 mg | EDP-305 2.5 mg
Number analyzed (Participants) | 54 | 52
h*ng/mL
  Day 1: number analyzed (Participants) | 19 | 19
  Day 1 | 1.48 (174) | 3.77 (112)
  Week 12: number analyzed (Participants) | 17 | 12
  Week 12 | 1.41 (187.01) | 3.81 (121.18)

23. Secondary Outcome: Cmax of EP-022572 on Day 1 and at Week 12
Description: The Cmax is the maximum observed plasma concentration, which was measured for EP-022572 (a metabolite of EDP-305) on Day 1 and Week 12 for the samples collected according to the intensive sampling scheme for the participants in the PK Population.
Time Frame: Predose and 2, 6, and 8 hours postdose on Day 1 and on Day 84 (Week 12)
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | EDP-305 1 mg | EDP-305 2.5 mg
Number analyzed (Participants) | 54 | 52
ng/mL
  Day 1: number analyzed (Participants) | 19 | 19
  Day 1 | 0.234 (1942) | 0.571 (212)
  Week 12: number analyzed (Participants) | 17 | 13
  Week 12 | 0.214 (2863) | 0.556 (212)

24. Secondary Outcome: Tmax of EP-022572 on Day 1 and at Week 12
Description: The Tmax was measured for EP-022572 (a metabolite of EDP-305) on Day 1 and at Week 12 for the samples collected according to the intensive sampling scheme for the participants in the PK Population.
Time Frame: Predose and 2, 6, and 8 hours postdose on Day 1 and on Day 84 (Week 12)
Population: as for outcome 17
Measure: Median (Full Range); unit: h
Arm/Group | EDP-305 1 mg | EDP-305 2.5 mg
Number analyzed (Participants) | 54 | 52
h
  Day 1: number analyzed (Participants) | 19 | 19
  Day 1 | 6.00 [2.00 to 8.07] | 6.00 [2.00 to 8.00]
  Week 12: number analyzed (Participants) | 17 | 13
  Week 12 | 6.00 [0.00 to 8.00] | 2.05 [0.00 to 8.18]

25. Secondary Outcome: AUC(Last) of EP-022572 on Day 1 and at Week 12
Description: AUC(last) is defined as the area under the plasma concentration-time curve from time zero to time the last quantifiable concentration, computed using the linear up/log down trapezoidal rule. AUC(last) was computed for EP-022572 (a metabolite of EDP-305) on Day 1 and Week 12 for the samples collected according to the intensive sampling scheme for the participants in the PK Population.
Time Frame: Predose and 2, 6, and 8 hours postdose on Day 1 and on Day 84 (Week 12)
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | EDP-305 1 mg | EDP-305 2.5 mg
Number analyzed (Participants) | 54 | 52
h*ng/mL
  Day 1: number analyzed (Participants) | 19 | 19
  Day 1 | 1.06 (220) | 2.92 (114)
  Week 12: number analyzed (Participants) | 17 | 12
  Week 12 | 1.13 (212) | 3.19 (116)

26. Secondary Outcome: Cmax of EP-022679 on Day 1 and at Week 12
Description: The Cmax is the maximum observed plasma concentration, which was measured for EP-022679 (a metabolite of EDP-305) on Day 1 and Week 12 for the samples collected according to the intensive sampling scheme for the participants in the PK Population.
Time Frame: Predose and 2, 6, and 8 hours postdose on Day 1 and on Day 84 (Week 12)
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | EDP-305 1 mg | EDP-305 2.5 mg
Number analyzed (Participants) | 54 | 52
ng/mL
  Day 1: number analyzed (Participants) | 19 | 19
  Day 1 | 0.574 (321) | 1.28 (167)
  Week 12: number analyzed (Participants) | 17 | 13
  Week 12 | 1.41 (117) | 3.85 (122)

27. Secondary Outcome: Tmax of EP-022679 on Day 1 and at Week 12
Description: The Tmax was measured for EP-022679 (a metabolite of EDP-305) on Day 1 and at Week 12 for the samples collected according to the intensive sampling scheme for the participants in the PK Population.
Time Frame: Predose and 2, 6, and 8 hours postdose on Day 1 and on Day 84 (Week 12)
Population: as for outcome 17
Measure: Median (Full Range); unit: h
Arm/Group | EDP-305 1 mg | EDP-305 2.5 mg
Number analyzed (Participants) | 54 | 52
h
  Day 1: number analyzed (Participants) | 19 | 19
  Day 1 | 8.00 [5.88 to 8.00] | 8.00 [6.00 to 8.25]
  Week 12: number analyzed (Participants) | 17 | 13
  Week 12 | 6.03 [0.00 to 8.00] | 6.00 [0.00 to 8.18]

28. Secondary Outcome: AUC(Last) of EP-022679 on Day 1 and at Week 12
Description: AUC(last) is defined as the area under the plasma concentration-time curve from time zero to time the last quantifiable concentration, computed using the linear up/log down trapezoidal rule. AUC(last) was computed for EP-022679 (a metabolite of EDP-305) on Day 1 and Week 12 for the samples collected according to the intensive sampling scheme for the participants in the PK Population.
Time Frame: Predose and 2, 6, and 8 hours postdose on Day 1 and on Day 84 (Week 12)
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | EDP-305 1 mg | EDP-305 2.5 mg
Number analyzed (Participants) | 54 | 52
h*ng/mL
  Day 1: number analyzed (Participants) | 19 | 19
  Day 1 | 2.32 (137.54) | 5.09 (117)
  Week 12: number analyzed (Participants) | 17 | 12
  Week 12 | 7.14 (113) | 22.5 (104)

29. Secondary Outcome: Mean Change From Baseline in Body Weight at Week 12
Description: Body weight was measured at specific timepoints for the participants. Baseline refers to the last non-missing value collected prior to the first dose of study treatment. Mean change was defined as the mean value at Week 12 minus the mean value at baseline.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | Placebo | EDP-305 1 mg | EDP-305 2.5 mg
Number analyzed (Participants) | 20 | 49 | 38
kilograms (kg) | -0.877 (2.8100) | -1.440 (2.7984) | -2.114 (3.2829)
Statistical Analysis 1: Comparison: Placebo vs EDP-305 2.5 mg; Test type: Superiority; p = 0.1120, ANCOVA; LS mean difference = 1.356, 95% CI 2-sided [-0.322 to 3.034]
Statistical Analysis 2: Comparison: Placebo vs EDP-305 1 mg; Test type: Superiority; p = 0.4229, ANCOVA; LS mean difference = 0.647, 95% CI 2-sided [-0.947 to 2.240]
Statistical Analysis 3: Comparison: EDP-305 1 mg vs EDP-305 2.5 mg; Test type: Superiority; p = 0.2764, ANCOVA; LS mean difference = 0.710, 95% CI 2-sided [-0.577 to 1.996]

30. Secondary Outcome: Mean Change From Baseline in Waist to Hip (WTH) Ratio at Week 12
Description: The WTH ratio is calculated as the ratio of waist to hip circumference, which was measured at specific timepoints. Baseline refers to the last non-missing value collected prior to the first dose of study treatment. Mean change was defined as the mean value at Week 12 minus the mean value at baseline.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Placebo | EDP-305 1 mg | EDP-305 2.5 mg
Number analyzed (Participants) | 19 | 49 | 38
ratio | 0.013 (0.0729) | -0.007 (0.0477) | 0.014 (0.0509)
Statistical Analysis 1: Comparison: Placebo vs EDP-305 2.5 mg; Test type: Superiority; p = 0.5606, ANCOVA; LS mean difference = 0.008, 95% CI 2-sided [-0.020 to 0.037]
Statistical Analysis 2: Comparison: Placebo vs EDP-305 1 mg; Test type: Superiority; p = 0.1002, ANCOVA; LS mean difference = 0.023, 95% CI 2-sided [-0.004 to 0.050]
Statistical Analysis 3: Comparison: EDP-305 1 mg vs EDP-305 2.5 mg; Test type: Superiority; p = 0.2002, ANCOVA; LS mean difference = -0.014, 95% CI 2-sided [-0.036 to 0.008]

31. Secondary Outcome: Mean Change From Baseline in Fibroblast Growth Factor 19 (FGF19) by Nominal Timepoint (Intensive Pharmacodynamic [PD] Samples) at Week 12
Description: Blood samples were collected according to the intensive sampling scheme at specific timepoints to assess the PD marker: FGF19. Baseline refers to the last non-missing predose value collected prior to the most recent dose of study treatment. Mean change was defined as the mean value at Week 12 minus the mean value at baseline.
Time Frame: Predose and 2, 6, and 8 hours postdose on Day 1 and Day 84 (Week 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nanogram per liter (ng/L)
Arm/Group | Placebo | EDP-305 1 mg | EDP-305 2.5 mg
Number analyzed (Participants) | 8 | 18 | 14
nanogram per liter (ng/L) | 159.98 (165.245) | 410.00 (260.223) | 607.12 (891.553)
Statistical Analysis 1: Comparison: Placebo vs EDP-305 2.5 mg; Test type: Superiority; p = 0.7014, ANCOVA; LS mean difference = -178.787, 95% CI 2-sided [-1098.454 to 740.880]
Statistical Analysis 2: Comparison: Placebo vs EDP-305 1 mg; Test type: Superiority; p = 0.9070, ANCOVA; LS mean difference = 52.307, 95% CI 2-sided [-830.934 to 935.547]
Statistical Analysis 3: Comparison: EDP-305 1 mg vs EDP-305 2.5 mg; Test type: Superiority; p = 0.5360, ANCOVA; LS mean difference = -231.094, 95% CI 2-sided [-967.273 to 505.086]

32. Secondary Outcome: Mean Change From Baseline in FGF19 by Bin Timepoint (Sparse PD Samples) at Week 12
Description: Blood samples were collected according to the sparse sampling scheme at specific timepoints to assess the PD marker: FGF19. Baseline refers to the last non-missing predose value collected prior to the most recent dose of study treatment. Mean change was defined as the mean value at Week 12 minus the mean value at baseline.
Time Frame: Predose and two samples postdose (first sample between 1 to 3 hours postdose and second sample 1 hour later than fist sample) on Day 1 and Day 84 (Week 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Placebo | EDP-305 1 mg | EDP-305 2.5 mg
Number analyzed (Participants) | 9 | 23 | 17
ng/L | 33.51 (155.744) | 46.04 (88.662) | 813.29 (3200.567)
Statistical Analysis 1: Comparison: Placebo vs EDP-305 2.5 mg; Test type: Superiority; p = 0.2985, ANCOVA; LS mean difference = -753.153, 95% CI 2-sided [-2183.920 to 677.614]
Statistical Analysis 2: Comparison: Placebo vs EDP-305 1 mg; Test type: Superiority; p = 0.8413, ANCOVA; LS mean difference = 139.107, 95% CI 2-sided [-1236.689 to 1514.902]
Statistical Analysis 3: Comparison: EDP-305 1 mg vs EDP-305 2.5 mg; Test type: Superiority; p = 0.1168, ANCOVA; LS mean difference = -892.260, 95% CI 2-sided [-2011.705 to 227.186]

33. Secondary Outcome: Mean Change From Baseline in 7a-Hydroxy-4-Cholestene-3-One (C4) by Nominal Timepoint (Intensive PD Samples) at Week 12
Description: Blood samples were collected according to the intensive sampling scheme at specific timepoints to assess the PD marker: C4. Baseline refers to the last non-missing predose value collected prior to the most recent dose of study treatment. Mean change was defined as the mean value at Week 12 minus the mean value at baseline.
Time Frame: Predose and 2, 6, and 8 hours postdose on Day 1 and Day 84 (Week 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | EDP-305 1 mg | EDP-305 2.5 mg
Number analyzed (Participants) | 8 | 17 | 14
ng/mL | -9.484 (20.6295) | -36.783 (24.6560) | -40.567 (20.9260)
Statistical Analysis 1: Comparison: Placebo vs EDP-305 2.5 mg; Test type: Superiority; p < 0.0001, ANCOVA; LS mean difference = 33.491, 95% CI 2-sided [17.984 to 48.998]
Statistical Analysis 2: Comparison: Placebo vs EDP-305 1 mg; Test type: Superiority; p < 0.0001, ANCOVA; LS mean difference = 30.814, 95% CI 2-sided [15.802 to 45.825]
Statistical Analysis 3: Comparison: EDP-305 1 mg vs EDP-305 2.5 mg; Test type: Superiority; p = 0.6757, ANCOVA; LS mean difference = 2.677, 95% CI 2-sided [-9.946 to 15.300]

34. Secondary Outcome: Mean Change From Baseline in C4 by Bin Timepoint (Sparse PD Samples) at Week 12
Description: Blood samples were collected according to the sparse sampling scheme at specific timepoints to assess the PD marker: C4. Baseline refers to the last non-missing predose value collected prior to the most recent dose of study treatment. Mean change was defined as the mean value at Week 12 minus the mean value at baseline.
Time Frame: as for outcome 32
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | EDP-305 1 mg | EDP-305 2.5 mg
Number analyzed (Participants) | 9 | 25 | 18
ng/mL | -5.242 (30.5321) | -13.500 (26.2458) | -23.773 (20.7045)
Statistical Analysis 1: Comparison: Placebo vs EDP-305 2.5 mg; Test type: Superiority; p = 0.0134, ANCOVA; LS mean difference = 21.300, 95% CI 2-sided [4.533 to 38.067]
Statistical Analysis 2: Comparison: Placebo vs EDP-305 1 mg; Test type: Superiority; p = 0.4686, ANCOVA; LS mean difference = 5.847, 95% CI 2-sided [-10.116 to 21.811]
Statistical Analysis 3: Comparison: EDP-305 1 mg vs EDP-305 2.5 mg; Test type: Superiority; p = 0.0181, ANCOVA; LS mean difference = 15.453, 95% CI 2-sided [2.699 to 28.206]

35. Secondary Outcome: Mean Change From Baseline in Bile Acid (BA) by Nominal Timepoint (Intensive PD Samples) at Week 12
Description: Blood samples were collected according to the intensive sampling scheme at specific timepoints to assess the PD marker: BA. Baseline refers to the last non-missing predose value collected prior to the most recent dose of study treatment. Mean change was defined as the mean value at Week 12 minus the mean value at baseline.
Time Frame: Predose and 2, 6, and 8 hours postdose on Day 1 and Day 84 (Week 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: micromoles per liter (μmol/L)
Arm/Group | Placebo | EDP-305 1 mg | EDP-305 2.5 mg
Number analyzed (Participants) | 7 | 18 | 14
micromoles per liter (μmol/L) | 4.47 (3.668) | 2.16 (5.507) | 0.14 (3.125)
Statistical Analysis 1: Comparison: Placebo vs EDP-305 2.5 mg; Test type: Superiority; p = 0.0557, ANCOVA; LS mean difference = 4.324, 95% CI 2-sided [-0.108 to 8.756]
Statistical Analysis 2: Comparison: Placebo vs EDP-305 1 mg; Test type: Superiority; p = 0.2867, ANCOVA; LS mean difference = 2.305, 95% CI 2-sided [-1.955 to 6.566]
Statistical Analysis 3: Comparison: EDP-305 1 mg vs EDP-305 2.5 mg; Test type: Superiority; p = 0.2437, ANCOVA; LS mean difference = 2.019, 95% CI 2-sided [-1.390 to 5.429]

36. Secondary Outcome: Mean Change From Baseline in BA by Bin Timepoint (Sparse PD Samples) at Week 12
Description: Blood samples were collected according to the sparse sampling scheme at specific timepoints to assess the PD marker: BA. Baseline refers to the last non-missing predose value collected prior to the most recent dose of study treatment. Mean change was defined as the mean value at Week 12 minus the mean value at baseline.
Time Frame: as for outcome 32
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Placebo | EDP-305 1 mg | EDP-305 2.5 mg
Number analyzed (Participants) | 9 | 25 | 17
μmol/L | 0.77 (5.789) | -0.11 (2.783) | 0.74 (4.091)
Statistical Analysis 1: Comparison: Placebo vs EDP-305 2.5 mg; Test type: Superiority; p = 0.9913, ANCOVA; LS mean difference = 0.019, 95% CI 2-sided [-3.491 to 3.530]
Statistical Analysis 2: Comparison: Placebo vs EDP-305 1 mg; Test type: Superiority; p = 0.5530, ANCOVA; LS mean difference = 0.995, 95% CI 2-sided [-2.323 to 4.314]
Statistical Analysis 3: Comparison: EDP-305 1 mg vs EDP-305 2.5 mg; Test type: Superiority; p = 0.4729, ANCOVA; LS mean difference = -0.976, 95% CI 2-sided [-3.665 to 1.713]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were reported from the date of signing the consent form to the date of completion of the participant's end of the study visit (Week 16). Ongoing AEs were followed beyond the end of the study visit at the discretion of the investigator.
Description: Treatment-emergent adverse events were summarized for the Safety Population, which included all the randomized participants who received at least one dose of the study treatment.
Arm/Group | Placebo | EDP-305 1 mg | EDP-305 2.5 mg
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/55 | 0/53
Serious Adverse Events (participants affected / at risk) | 1/24 | 1/55 | 0/53
Other Adverse Events (participants affected / at risk) | 8/24 | 17/55 | 32/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=24) | EDP-305 1 mg (N=55) | EDP-305 2.5 mg (N=53)
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=24) | EDP-305 1 mg (N=55) | EDP-305 2.5 mg (N=53)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 5 | 25
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 3
Nausea (Gastrointestinal disorders) | 1 | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 3
Vomiting (Gastrointestinal disorders) | 2 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 3 | 1
Headache (Nervous system disorders) | 2 | 2 | 2
Dizziness (Nervous system disorders) | 1 | 3 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 3 | 1
Fatigue (General disorders) | 2 | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-02-21): https://cdn.clinicaltrials.gov/large-docs/31/NCT03421431/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-05): https://cdn.clinicaltrials.gov/large-docs/31/NCT03421431/SAP_001.pdf